CLINICAL TRIAL: NCT00416520
Title: A Phase III, Randomised, Double-Blind, Multi-centre, Withdrawal Study Comparing MCI-196 Versus Placebo in Chronic Kidney Disease Stage V Subjects on Dialysis With Hyperphosphatemia
Brief Title: A Phase III, Multicentre, Double-Blind, Placebo-Controlled Withdrawal Study in Patients With Hyperphosphatemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MCI-196-E07
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Results first posted 2014-10-23 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Chronic Kidney Disease; Hyperphosphatemia
Keywords: Chronic Kidney Disease; Dialysis; Hyperphosphatemia; Phosphate binder
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperphosphatemia | interventions — cholebine; Sevelamer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: MCI-196 (Colestilan(INN), Colestimide(JAN), CHOLEBINE®)
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo
- 3 (Active Comparator)
  Interventions: Drug: Another phosphate binder (Sevelamer)

INTERVENTIONS:
Drug: MCI-196 (Colestilan(INN), Colestimide(JAN), CHOLEBINE®) — 3g to 15g/day (3 times a day), Tablet, 12 weeks of flexible dose and 4 weeks of double blind
  Arms: 1
Drug: Placebo — 3g to 15g/day (3 times a day), Tablet, 4 weeks of double blind
  Arms: 2
Drug: Another phosphate binder (Sevelamer) — Current approved dosing recommendations for 12 weeks
  Arms: 3

SUMMARY:
This is a phase III multi-centre study in three periods: the first period is a phosphate binder washout for 4 weeks, the second period is an open-label, randomised, parallel group, flexible dose, the third period is a placebo-controlled withdrawal comparing MCI-196 with placebo for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or over
* Clinically stable haemodialysis or peritoneal dialysis
* Stable phosphate control
* On a stabilised phosphorus diet
* Female and of child-bearing potential have a negative serum pregnancy test.
* Male subjects must agree to use appropriate contraception.

Exclusion Criteria:

* Current clinically significant medical comorbidities, which may substantially compromise subject safety, or expose them to undue risk, or interfere significantly with study procedures and which, in the opinion of the Investigator, makes the subject unsuitable for inclusion in the study.
* Body Mass Index (BMI) <=16.0 kg/m2 or >=40.0 kg/m2
* A current or history of significant gastrointestinal motility problems
* A positive test for HIV 1 and 2 antibodies
* A history of substance or alcohol abuse within the last year.
* Seizure disorders
* A history of drug or other allergy
* A temporary catheter as a vascular access
* Participated in a clinical study with any experimental medication in the last 30 days or an experimental biological product within the last 90 days prior to signing of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2007-06; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Professor, Principal Investigator — Information at Mitsubishi Pharma Europe
Locations (68):
- Australia (6):
  - Adelaide
  - Nedlands
  - Parkville
  - St Leonards
  - Sydney
  - Woolloongabba
- Graz, Austria
- Czechia (6):
  - Frýdek-Místek
  - HradecKralove
  - Ostrava
  - Prague
  - Tábor
  - Ústí nad Labem
- France (3):
  - Bordeaux
  - Montpelier
  - Paris
- Germany (14):
  - Aachen
  - Aschaffenburg
  - Coburg
  - Coesfeld
  - Darmstadt
  - Dieburg
  - Dortmund
  - Düsseldorf
  - Hamburg
  - Homberg (Efze)
  - Langen
  - Mannheim-Kafertal
  - München
  - Potsdam-Babelsberg
- Hungary (4):
  - Baja
  - Budapest
  - Kisvárda
  - Veszprém
- Italy (9):
  - Biella
  - Como
  - Cremona
  - Lecco
  - Livorno
  - Milan
  - Pavia
  - Perugia
  - Rome
- Poland (15):
  - Ciechanów
  - Częstochowa
  - Gdansk
  - Krakow
  - Lodz
  - Lublin
  - Oświęcim
  - Pabianice
  - Rybnik
  - Sokołów Podlaski
  - Starogard Gdański
  - Warsaw
  - Wejherowo
  - Zgierz
  - Zielona Góra
- South Africa (5):
  - Cape Town
  - Durban
  - Gauteng
  - Johannesburg
  - Port Elizabeth
- Spain (3):
  - Barcelona
  - Oviedo
  - Seville
- United Kingdom (2):
  - Glasgow
  - Stevenage

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086

RESULTS

PARTICIPANT FLOW:
Groups:
- MCI-196 (Open-label Period): 3, 6, 9, 12, or 15g/day as titrated
  * There was a gap of 3 subjects between "STARTED" and "Overall Number of Baseline Participants".
  * Two subjects were randomised to receive MCI-196, but did not take study medication. These 2 subjects were excluded from "Baseline Participants" of MCI-196 group.
  * In addition, one subject (A) was randomised to receive MCI-196, but took sevelamer instead. This subject was counted as MCI-196 group for "STARTED" but counted as Sevelamer group for "Baseline Participants".
- Sevelamer (Open-label Period): 2.4, 4.8, 7.2, 9.6, or 12.0g/day as titrated
  * There was a gap of 2 subjects between "STARTED" and "Overall Number of Baseline Participants".
  * Three subjects in Sevelamer group were randomised in error and did not take any study medication. These 3 subjects were excluded from "Baseline Participants" of Sevelamer group.
  * However, one subject (A) was randomised to receive MCI-196, but took sevelamer instead. This subject was counted as MCI-196 group for "STARTED" but counted as Sevelamer group for "Baseline Participants".
- MCI-196 (Placebo-controlled Withdrawal Period): dose level at the end of dose titration in the flexible dose period
- Placebo (Placebo-controlled Withdrawal Period): dose level at the end of dose titration in the flexible dose period
  There was a gap of 1 subject between "STARTED" and "Overall Number of Baseline Participants" One subject did not take any study medication and excluded from "Baseline Participants".
Period: Open-label Period
Arm/Group | MCI-196 (Open-label Period) | Sevelamer (Open-label Period) | MCI-196 (Placebo-controlled Withdrawal Period) | Placebo (Placebo-controlled Withdrawal Period)
Started | 165 | 171 | 0 | 0
Completed | 105 | 139 | 0 | 0
Not Completed | 60 | 32 | 0 | 0
Not completed — Adverse Event | 28 | 10 | 0 | 0
Not completed — Death | 2 | 1 | 0 | 0
Not completed — Lack of Efficacy | 8 | 1 | 0 | 0
Not completed — Protocol Violation | 3 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 16 | 5 | 0 | 0
Not completed — Other Reasons | 3 | 12 | 0 | 0
Period: Placebo-controlled Withdrawal Period
Arm/Group | MCI-196 (Open-label Period) | Sevelamer (Open-label Period) | MCI-196 (Placebo-controlled Withdrawal Period) | Placebo (Placebo-controlled Withdrawal Period)
Started | 0 | 0 | 50 | 54
Completed | 0 | 0 | 49 | 49
Not Completed | 0 | 0 | 1 | 5
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 3
Not completed — Protocol Violation | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MCI-196 (Open-label Period) | Sevelamer (Open-label Period) | Total
Number analyzed (Participants) | 162 | 169 | 331
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (14.7) | 59.5 (13.8) | 58.0 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 72 | 126
  Male | 108 | 97 | 205

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Phosphorus Levels From Week 12 to Week 16 (LOCF) (ITT2)
Description: ITT2 population included all re-randomised subjects who completed 12 weeks in the MCI-196 treatment group and received at least 1 dose of study medication in the placebo-controlled withdrawal period and had at least 1 central serum phosphorus value after 12 weeks.
Time Frame: week16 minus week12
Population: ITT2 population included all re-randomised subjects who completed 12 weeks in the MCI-196 treatment group and received at least 1 dose of study medication in the placebo-controlled withdrawal period and had at least 1 central serum phosphorus value after 12 weeks.
Measure: Mean (Standard Deviation); unit: mg / dL
Groups:
- Placebo (Placebo-controlled Withdrawal Period): dose level at the end of dose titration in the flexible dose period
Arm/Group | MCI-196 (Placebo-controlled Withdrawal Period) | Placebo (Placebo-controlled Withdrawal Period)
Number analyzed (Participants) | 50 | 53
mg / dL | -0.24 (1.46) | 1.27 (1.48)

2. Secondary Outcome: Change in Serum Phosphorus Levels From Baseline to Week 12 (LOCF) (ITT1)
Description: ITT1 population included all subjects who received a randomisation number (at Week 0), took at least 1 dose of study medication and had at least 1 central serum phosphorus value after the start of study medication.
Time Frame: week12 minus week0
Population: ITT1 population included all subjects who received a randomisation number (at Week 0), took at least 1 dose of study medication and had at least 1 central serum phosphorus value after the start of study medication.
Measure: Mean (Standard Deviation); unit: mg / dL
Groups:
- MCI-196 (Open-label Period): 3, 6, 9, 12, or 15g/day as titrated
- Sevelamer (Open-label Period): 2.4, 4.8, 7.2, 9.6, or 12.0g/day as titrated
Arm/Group | MCI-196 (Open-label Period) | Sevelamer (Open-label Period)
Number analyzed (Participants) | 160 | 167
mg / dL | -1.12 (1.63) | -2.16 (1.55)

ADVERSE EVENTS:
Groups:
- MCI-196 (Placebo-Controlled Period); Placebo (Placebo-Controlled Period): dose level at the end of dose titration in the flexible dose period
Arm/Group | MCI-196 (Open-label Period) | Sevelamer (Open-label Period) | MCI-196 (Placebo-Controlled Period) | Placebo (Placebo-Controlled Period)
Serious Adverse Events (participants affected / at risk) | 26/162 | 25/169 | 2/50 | 3/53
Other Adverse Events (participants affected / at risk) | 126/162 | 113/169 | 20/50 | 23/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MCI-196 (Open-label Period) (N=162) | Sevelamer (Open-label Period) (N=169) | MCI-196 (Placebo-Controlled Period) (N=50) | Placebo (Placebo-Controlled Period) (N=53)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 2 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiovascular insufficiency (Cardiac disorders) | 0 | 1 | 0 | 0
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 1 | 0 | 0
Coronary artery insufficiency (Cardiac disorders) | 0 | 1 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 3 | 0 | 0 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hernia (General disorders) | 0 | 1 | 0 | 0
Impaired healing (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1 | 1 | 0
Catheter sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Arteriogram coronary (Investigations) | 0 | 2 | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Genital haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Cataract operation (Surgical and medical procedures) | 1 | 0 | 0 | 0
Coronary arterial stent insertion (Surgical and medical procedures) | 0 | 1 | 0 | 0
Renal transplant (Surgical and medical procedures) | 1 | 1 | 0 | 0
Toe amputation (Surgical and medical procedures) | 1 | 0 | 0 | 0
Circulatory collapse (Vascular disorders) | 1 | 0 | 0 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Dialysis device complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MCI-196 (Open-label Period) (N=162) | Sevelamer (Open-label Period) (N=169) | MCI-196 (Placebo-Controlled Period) (N=50) | Placebo (Placebo-Controlled Period) (N=53)
Anaemia (Blood and lymphatic system disorders) | 6 | 6 | 0 | 2
Angina pectoris (Cardiac disorders) | 2 | 2 | 0 | 0
Hyperparathyroidism (Endocrine disorders) | 2 | 1 | 0 | 0
Hyperparathyroidism secondary (Endocrine disorders) | 2 | 1 | 0 | 1
Eye haemorrhage (Eye disorders) | 0 | 2 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 8 | 4 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 10 | 8 | 1 | 0
Constipation (Gastrointestinal disorders) | 13 | 11 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 21 | 16 | 2 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 13 | 6 | 0 | 1
Eructation (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 4 | 2 | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 2 | 2 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 15 | 12 | 0 | 1
Vomiting (Gastrointestinal disorders) | 27 | 9 | 1 | 0
Asthenia (General disorders) | 2 | 0 | 0 | 0
Catheter site erythema (General disorders) | 0 | 2 | 0 | 0
Catheter site pain (General disorders) | 2 | 0 | 0 | 0
Chest pain (General disorders) | 2 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 0 | 0 | 0
Oedema peripheral (General disorders) | 2 | 1 | 2 | 0
Pyrexia (General disorders) | 5 | 2 | 0 | 0
Bronchitis (Infections and infestations) | 5 | 3 | 2 | 1
Bronchopneumonia (Infections and infestations) | 2 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 2 | 0 | 0
Cystitis (Infections and infestations) | 0 | 3 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 2 | 1 | 0
Influenza (Infections and infestations) | 1 | 4 | 0 | 0
Nasopharyngitis (Infections and infestations) | 8 | 7 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 5 | 0 | 0
Respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 0 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 4 | 0 | 0 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 2 | 2 | 0 | 0
Haemodialysis-induced symptom (Injury, poisoning and procedural complications) | 6 | 9 | 3 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0
Procedural hypertension (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 3 | 7 | 0 | 0
Blood parathyroid hormone increased (Investigations) | 1 | 3 | 1 | 0
C-reactive protein increased (Investigations) | 2 | 2 | 1 | 1
Electrocardiogram QT interval abnormal (Investigations) | 3 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 3 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 2 | 1 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 8 | 6 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 4 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 4 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 1 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 5 | 1 | 0
Headache (Nervous system disorders) | 6 | 5 | 1 | 1
Hypotonia (Nervous system disorders) | 1 | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 2 | 0 | 2
Sleep disorder (Psychiatric disorders) | 2 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 5 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0
Renal transplant (Surgical and medical procedures) | 2 | 4 | 0 | 0
Hypertension (Vascular disorders) | 12 | 12 | 1 | 1
Hypotension (Vascular disorders) | 1 | 6 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Spontaneous haematoma (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 1
Catheter site infection (Infections and infestations) | 0 | 1 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 2 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Eschar (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 1
Vitamin D decreased (Investigations) | 0 | 1 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Restless legs syndrome (Nervous system disorders) | 0 | 1 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other